CLINICAL TRIAL: NCT00642629
Title: A Randomized, Double-blind, Placebo-controlled Clinical Study of the Oral IL-12/23 Inhibitor, STA-5326 Mesylate, Administered to Patients With Rheumatoid Arthritis to Determine Safety, Tolerability, Pharmacokinetic and Synovial Tissue Outcomes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5326-09
Record Dates: First submitted 2008-03-20; First posted 2008-03-25 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Active, Moderate to Severe Rheumatoid Arthritis
MeSH Terms: conditions — Motor Activity | interventions — apilimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): STA-5326 mesylate
  Interventions: Drug: STA 5326 mesylate
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: STA 5326 mesylate — STA 5326 mesylate 100mg taken orally twice a day for 8 weeks with the option to continue at the same dose and frequency for an additional 4 weeks.
  Arms: 1
Drug: Placebo — Placebo taken orally twice a day for 8 weeks with the option to continue at the same dose and frequency for an additional 4 weeks.
  Arms: 2

SUMMARY:
It is not fully clear how rheumatoid arthritis originates and develops, but it is understood that multiple genetic and environmental factors interact to trigger its onset. The immune system attacks the joint synovium, which damages the cartilage and bone in the joint by increasing the number of inflammatory cells and forming new blood vessels in the joint space. STA-5326 mesylate inhibits the production of IL-12 and IL-23 and therefore may inhibit Th-1 cytokine production. A reduction in the Th-1 response has the potential to minimize or eliminate joint damage caused by the immune response in rheumatoid arthritis. This study is designed to assess whether the proposed mechanism of action is associated with a reduction in inflammation in the synovium of patients who have rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older.
* Has a diagnosis of RA in conformance with the American College of Rheumatology (ACR) criteria for at least 6 months.
* Has at least one knee, wrist, or ankle that has active synovitis and is amenable to arthroscopic procedures for the acquisition of synovial tissue via biopsy.
* Must be taking methotrexate for a minimum of 4 months prior to Day 1, with a stable dose regimen for at least 2 months, and
* have plans to remain on the stable dose regimen of methotrexate for the duration of this study.
* If female of childbearing potential, must be neither pregnant nor breast feeding, and
* must have a negative pregnancy test (serum β-hCG) within 1 week of Day 1. Must be willing to use "double-barrier" contraception methods for the duration of the study.

Exclusion Criteria:

* Is taking any disease-modifying anti-rheumatic drug (DMARD) other than MTX concomitantly or within 1 month prior to Day 1.
* A positive (≥10 mm) tuberculin (PPD) skin test, unless the patient has had prior BCG immunization or has received prior suppressive treatment such as 1 year of INH.
* Has received any investigational drug or experimental procedure for the treatment of RA within 3 months of Day 1 for a biologic compound or within 1 month of Day 1 for a non-biologic compound.
* Has any clinically significant disease (e.g., renal, hepatic, neurological, cardiovascular, pulmonary, endocrine, psychiatric, hematologic, urologic, or other acute or chronic illness) that, in the opinion of the investigator, would make the patient an unsuitable candidate for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2005-12

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Krausz S, Boumans MJ, Gerlag DM, Lufkin J, van Kuijk AW, Bakker A, de Boer M, Lodde BM, Reedquist KA, Jacobson EW, O'Meara M, Tak PP. Brief report: a phase IIa, randomized, double-blind, placebo-controlled trial of apilimod mesylate, an interleukin-12/interleukin-23 inhibitor, in patients with rheumatoid arthritis. Arthritis Rheum. 2012 Jun;64(6):1750-5. doi: 10.1002/art.34339. Epub 2011 Dec 14. PMID 22170479